CLINICAL TRIAL: NCT01190150
Title: Randomized, 2-way Crossover, Pharmacokinetic Study of Lysteda (Xanodyne Modified-Immediate Release Tranexamic Acid) Tablets at 2 Doses in Fasting Adolescent Females With Evidence of Heavy Menstrual Bleeding
Brief Title: Lysteda Pediatric Research Equity Act (PREA) Pharmacokinetic Study in Adolescent Females With Heavy Menstrual Bleeding
Acronym: PREA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: FE999304 CS01
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Results first posted 2012-07-03 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Menorrhagia
Keywords: Cyclic Heavy Menstrual Bleed; Menorraghia
MeSH Terms: conditions — Menorrhagia | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.65 g / 1.3 g tranexamic acid (Experimental): Participants received a single dose of 0.65 g tranexamic acid on Day 1 and a single dose of 1.3 g tranexamic acid on Day 8.
  Interventions: Drug: tranexamic acid
- 1.3 g / 0.65 g tranexamic acid (Experimental): Participants received a single dose of 1.3 g tranexamic acid on Day 1 and a single dose of 0.65 g tranexamic acid on Day 8.
  Interventions: Drug: tranexamic acid

INTERVENTIONS:
Drug: tranexamic acid — Either one or two modified-immediate release tranexamic acid tablets (0.65 g each) taken orally, administered with 240 mL of water, as a single dose, at approximately 8 AM.
  Other Names: Lysteda; modified-immediate release tranexamic acid

SUMMARY:
This is a Phase 4, randomized, 2-way crossover, pharmacokinetic study of Lysteda (tranexamic acid) tablets administered as single doses of 0.65 g and 1.3 g in fasting adolescent female subjects ages 12-16 years with heavy menstrual bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy non-smoking (for at least 3 months) adolescent females 12-16 years of age with a history of at least 1 year of cyclic heavy menstrual bleeding (HMB)
* Subjects must report regularly occurring menstrual periods ≤10 days in duration, with 21-45 days from the start of one period to the start of the next menstrual period
* Diagnosis of HMB based on the medical judgment of the Principal Investigator and will include the following criteria:

  1. Laboratory (including a bleeding disorders work-up) and Physical Findings;
  2. Limitations in Activities of Daily Living (ADL);
  3. Soiling, Staining and Clotting;
  4. Sanitary product usage and extent of MBL using a patient reported pictorial blood assessment chart (PBAC).
* Subjects should either be sexually inactive (abstinent) or be using one of the following acceptable birth control methods and agree to continue its use throughout the study:

  * copper intrauterine device (IUD) in place for at least 3 months;
  * barrier methods (condom, diaphragm) with spermicide for at least 1 month prior to the first dose and throughout the study.
* Negative pregnancy test results
* Subject's legally authorized representative (e.g., parent, guardian) must voluntarily sign a parental permission/informed consent form (ICF), and the subject must sign an assent, before the conduct of any study procedure

Exclusion Criteria:

* Breast-feeding, or a history of abortion in the last 6 months
* Known bleeding or coagulation disorders based on medical history and/or laboratory results
* Known systemic hematologic diseases (e.g., all types of sickle-cell disease, thalassemia of all types, multiple myeloma, hemolytic anemia)
* Clinical evidence of any significant chronic illness, including cardiovascular, renal, neurologic, hepatic, endocrine, gastric, central nervous system disease, any psychiatric illness which could affect the efficacy or safety of study medication
* Subjects treated with systemic steroids in the last 1 month or hormonal treatment in the last 3 months
* A history or presence of any drug abuse or alcohol abuse within the last 1 year
* History of subarachnoid hemorrhage.
* Active thromboembolic disease; history of thrombosis or thromboembolism, including retinal vein or artery occlusion; an intrinsic risk of thrombosis or thromboembolism
* Use of vaginal hormone products (rings, creams, and gels) within 4 weeks prior to screening. Use of oral estrogen-, progestin-, or selective estrogen receptor within 8 weeks prior to screening. Use of Lupron (3-month depot injection), estrogen pellet, or long-acting progestin injectables within 6 months prior to screening
* Subjects whose sitting blood pressure is less than 90/60 mmHg at screening
* Subjects whose pulse is lower than 50 b.p.m. at screening
* Subjects whose PR interval is >200 msec at screening and prior to dosing
* Subjects whose QTc interval >450 msec
* Subjects with positive tests for hepatitis B, C, or human immunodeficiency virus (HIV)

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Period: First Treatment
Arm/Group | 0.65 g / 1.3 g Tranexamic Acid | 1.3 g / 0.65 g Tranexamic Acid
Started | 11 (Randomized, as well as Safety and PK populations) | 9 (Randomized, as well as Safety and PK populations)
Completed | 10 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout
Arm/Group | 0.65 g / 1.3 g Tranexamic Acid | 1.3 g / 0.65 g Tranexamic Acid
Started | 10 | 9
Completed | 10 | 7
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Difficulty in adherence | 0 | 1
Period: Second Treatment
Arm/Group | 0.65 g / 1.3 g Tranexamic Acid | 1.3 g / 0.65 g Tranexamic Acid
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.65 g / 1.3 g Tranexamic Acid | 1.3 g / 0.65 g Tranexamic Acid | Total
Number analyzed (Participants) | 11 | 9 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.13) | 14.3 (1.32) | 14.4 (1.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentrations Level (Cmax)
Description: Cmax is the maximum measured plasma concentration over the time-span specified.
Time Frame: Day 1 or Day 8 (before dosing and at the following times thereafter: 0.5, 0.75, 1, 2, 2.5, 3.0, 3.5, 4, 5, 6, 10, 14, and 24 hours post-dose)
Population: Plasma PK population includes all participants with at least one quantifiable PK concentration.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- 0.65 g Tranexamic Acid: Participants were treated with a single dose of 0.65 g tranexamic acid.
- 1.3 g Tranexamic Acid: Participants were treated with a single dose of 1.3 g tranexamic acid.
Arm/Group | 0.65 g Tranexamic Acid | 1.3 g Tranexamic Acid
Number analyzed (Participants) | 18 | 19
μg/mL | 6.9967 (2.08058) | 10.9868 (3.38910)

2. Primary Outcome: Dose-normalized Maximum Concentrations Level (Cmax)
Description: Cmax is the maximum measured plasma concentration over the time-span specified and normalized to the 1.3 g dose.
Time Frame: as for outcome 1
Population: Plasma PK population includes all participants with at least one quantifiable PK concentration.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 0.65 g Tranexamic Acid | 1.3 g Tranexamic Acid
Number analyzed (Participants) | 18 | 19
μg/mL | 13.9933 (4.16115) | 10.9868 (3.38910)

3. Primary Outcome: Time to Maximum Concentration Level (Tmax)
Description: Time of the maximum measured plasma concentration. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value.
Time Frame: as for outcome 1
Population: Plasma PK population includes all participants with at least one quantifiable PK concentration.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 0.65 g Tranexamic Acid | 1.3 g Tranexamic Acid
Number analyzed (Participants) | 18 | 19
hours | 3.17 (0.642) | 3.11 (0.679)

4. Primary Outcome: Area Under the Concentration Versus Time Curve From 0 to the Last Time Point (AUC0-t)
Description: The area under the plasma concentration versus time curve, from time 0 to the last measurable concentration, as calculated by the linear trapezoidal method.
Time Frame: as for outcome 1
Population: Plasma PK population includes all participants with at least one quantifiable PK concentration.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | 0.65 g Tranexamic Acid | 1.3 g Tranexamic Acid
Number analyzed (Participants) | 18 | 19
μg*h/mL | 38.8067 (10.56742) | 56.7935 (19.27448)

5. Primary Outcome: Dose Normalized Area Under the Concentration Versus Time Curve From 0 to the Last Time Point (AUC0-t)
Description: The area under the plasma concentration versus time curve, from time 0 to the last measurable concentration normalized to the 1.3 g dose.
Time Frame: as for outcome 1
Population: Plasma PK population includes all participants with at least one quantifiable PK concentration.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | 0.65 g Tranexamic Acid | 1.3 g Tranexamic Acid
Number analyzed (Participants) | 18 | 19
μg*h/mL | 77.6134 (21.13483) | 56.7935 (19.27448)

6. Primary Outcome: Area Under the Concentration Versus Time Curve From 0 to Infinity (AUCinf)
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUCinf is calculated as the sum of AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: Plasma PK population including all participants with three or more non-zero plasma concentrations. One participant withdrew on Day 7 and did not meet the requisite samples required for this PK parameter.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | 0.65 g Tranexamic Acid | 1.3 g Tranexamic Acid
Number analyzed (Participants) | 18 | 18
μg*h/mL | 39.8016 (10.71237) | 61.2591 (15.45770)

7. Primary Outcome: Dose Normalized Area Under the Concentration Versus Time Curve From 0 to Infinity (AUCinf)
Description: Dose-normalized AUCinf is calculated as the sum of AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant, normalized to the 1.3 g dose.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | 0.65 g Tranexamic Acid | 1.3 g Tranexamic Acid
Number analyzed (Participants) | 18 | 18
μg*h/mL | 79.6032 (21.42474) | 61.2591 (15.45770)

8. Primary Outcome: The Ratio of AUC0-t to AUCinf
Description: Comparison of AUC0-t to AUCinf by creating a ratio.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio of AUC0-t / AUCinf
Arm/Group | 0.65 g Tranexamic Acid | 1.3 g Tranexamic Acid
Number analyzed (Participants) | 18 | 18
ratio of AUC0-t / AUCinf | 0.9741 (0.00862) | 0.9715 (0.01158)

9. Primary Outcome: Elimination Half-life (t ½)
Description: Apparent first-order terminal elimination half life
Time Frame: as for outcome 1
Population: Plasma PK population includes all participants with at least one quantifiable PK concentration.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 0.65 g Tranexamic Acid | 1.3 g Tranexamic Acid
Number analyzed (Participants) | 18 | 18
hours | 5.06 (1.194) | 5.42 (1.463)

10. Secondary Outcome: Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Treatment-emergent AEs are summarized by total participants with TEAEs, participants with serious TEAEs, participants with TEAEs deemed by the investigator to be related to treatment, and participants who experienced TEAEs that caused permanent discontinuation from the study.
Time Frame: Day 1 up to week 4
Population: The Safety Population consisted of all randomized participants who received at least one dose of tranexamic acid.
Measure: Number; unit: participants
Arm/Group | 0.65 g Tranexamic Acid | 1.3 g Tranexamic Acid
Number analyzed (Participants) | 18 | 19
participants
  Participants with TEAEs | 1 | 2
  Participants with serious TEAEs | 0 | 0
  Participants with treatment-related TEAEs | 0 | 1
  Participants with TEAEs causing discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to week 4
Arm/Group | 0.65 g Tranexamic Acid | 1.3 g Tranexamic Acid
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 1/18 | 2/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.65 g Tranexamic Acid (N=18) | 1.3 g Tranexamic Acid (N=19)
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.